CLINICAL TRIAL: NCT00069615
Title: DirecNet Pilot Study to Evaluate the GlucoWatch G2 Biographer in the Management of Type 1 Diabetes in Children
Brief Title: Pilot Study of the GlucoWatch G2 Biographer for the Management of Type 1 Diabetes in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: DirecNet 003; HD041890; HD041919-01; HD041908-01; HD041906-01; HD041918-01; HD041915
Record Dates: First submitted 2003-09-29; First posted 2003-09-30 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Mellitus, Insulin-Dependent
Keywords: Diabetes Mellitus, Insulin-Dependent; Type 1 Diabetes; Continuous Glucose Monitoring Devices; Electronic Data Collection
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Continuous Glucose Monitoring

INTERVENTIONS:
Device: GlucoWatch® G2™ Biographer (GW2B)
Device: Continuous Glucose Monitoring System™ (CGMS)

SUMMARY:
Devices such as the GlucoWatch G2 Biographer (GW2B), which constantly measure blood sugar levels, may improve the treatment of Type 1 diabetes mellitus in children. This study evaluated the GW2B when used by children in their homes.

DETAILED DESCRIPTION:
The proper role of the GW2B in the management of Type 1 diabetes in children has not been determined. As a prelude to a large-scale randomized clinical trial (RCT) to compare the effect on glycemic control, hypoglycemia, and quality of life of using a GW2B versus standard care, the DirecNet Study Group conducted a pilot study to assess the feasibility of the protocol planned for the RCT and to collect data on changes in HbA1c, frequency of hypoglycemia, frequency of skin reactions, and quality of life after using the GW2B for three months.

Fifteen children and adolescents with Type 1 diabetes participated in this study. Each patient was provided with a personal computer for weekly downloading of the GW2B and for completion of questionnaires regarding hypoglycemia and GW2B use. Participants received study telephone calls after 1, 2, and 4 weeks and every 4 weeks thereafter to review their diabetes management. Participants had a follow-up visit at Week 29. The Continuous Glucose Monitoring System was inserted at this visit to assess hypoglycemia over three days. A follow-up visit was performed at Week 30 to measure HbA1c and administer psychosocial questionnaires.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of Type 1 diabetes
* Duration of diabetes > 1 year
* Daily insulin therapy (pump or at least 2 injections/day)
* Stable insulin regimen; not expected to change administration modality within the next 3 months (e.g., injection user switching to pump)

Exclusion Criteria

* The presence of skin abnormalities or a significant medical disorder that in the judgment of the investigator will affect the wearing of the sensors or the completion of any aspect of the protocol.
* Prior use of a GWB prescribed for home use (Prior use of a GWB as part of a research study is allowable)
* The presence of any of the following diseases:

  * Asthma if treated with systemic or inhaled corticosteroids in the last 6 months
  * Cystic fibrosis
  * Other major illness that in the judgment of the investigator might interfere with the completion of the protocol
  * Adequately treated thyroid disease and celiac disease do not exclude
* Inpatient psychiatric treatment in the past 6 months for either the subject or the subject's primary care giver (i.e., parent or guardian).
* Current use of oral/inhaled glucocorticoids or other medications, which in the judgment of the investigator would be a contraindication to participation in the study.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15
Dates: Start 2003-02; Study Completion 2003-06

PRIMARY OUTCOMES:
Feasibility of using the GlucoWatch G2 Biographer
Feasibility of collecting data from home computers

CONTACTS AND LOCATIONS:
Overall Officials: William V Tamborlane, MD, Study Chair — Yale University
Locations (6):
- United States (6):
  - Division of Pediatric Endocrinology and Diabetes, Stanford University, Stanford, California
  - Barbara Davis Center for Childhood Diabetes, University of Colorado, Denver, Colorado
  - Department of Pediatrics, Yale University School of Medicine, New Haven, Connecticut
  - Nemours Children's Clinic, Jacksonville, Florida
  - Jaeb Center for Health Research, Tampa, Florida
  - Department of Pediatrics, University of Iowa Carver College of Medicine, Iowa City, Iowa

REFERENCES:
- [Background] Stuart Weinzimer, Katrina Ruedy, Jennifer Fisher, Linda Larson, Jennifer Block, Elizabeth Boland, Keisha Bird, and the Diabetes Research in Children Network (DirecNet) Study Group: Diabetes Research in Children Network (DirecNet) Outpatient Pilot Study to Evaluate the GlucoWatch G2 Biographer (GW2B) in the Management of Type 1 Diabetes (T1DM) in Children. Diabetes Technol Ther 2004; 6(2):280.
- [Background] Stuart Weinzimer, Katrina Ruedy, Linda Larson, Jennifer Block, Jennifer Fisher, Elizabeth Doyle, Keisha Bird, and the Diabetes Research in Children Network (DirecNet) Study Group: Diabetes Research in Children Network (DirecNet) Outpatient Pilot Study to Evaluate the Feasibility of Computer-Based Data Acquisition and Transmission. Pediatr Res 2004; 55 (4 Pt 2):138A.